CLINICAL TRIAL: NCT05167669
Title: Pain Relief in Patients With Symptomatic Bone Metastases: a Feasibility Pilot Study on Palliative Radiotherapy With Adjuvant Hyperthermia by Magnetic Resonance-guided Focused Ultrasound
Brief Title: Pain Relief in Symptomatic Bone Metastases With Adjuvant Hyperthermia MR Guided HIFU
Acronym: BM-RT-HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Boudabbous (Other)
Responsible Party: Sponsor-Investigator, Sana Boudabbous, MD PD HEAD OF MUSCULOSKELETAL UNITY- RADIOLOGY DIVISION- DIAGNOSIS DEPARTMENT, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02998
Record Dates: First submitted 2021-11-24; First posted 2021-12-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Bone Metastases; Radiotherapy; Pain; MRI
Keywords: BONE METASTASES, PAIN, MRI, HIFU, RADIOTHERAPY
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Number of participants: 10 patients with radiologically confirmed bone metastases and eligible for a course of palliative EBRT. Eligible patients will be mainly discussed and recruited in a dedicated tumor-board for bone metastases performed in a weekly basis at HUG.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prospective, interventional, single-center, feasibility pilot study. (Other): 10 patients with radiologically confirmed bone metastases and eligible for a course of palliative EBRT. Eligible patients will be mainly discussed and recruited in a dedicated tumor-board for bone metastases performed in a weekly basis at HUG.
  Interventions: Device: HIFU-MRI guided

INTERVENTIONS:
Device: HIFU-MRI guided — HIFU application under MRI guiding to deliver hypothermia to eligible bone metastases before clinical indicated radiotherapy

SUMMARY:
Metastatic disease to the bone is a common cause of pain. External beam radiation therapy (EBRT) is the standard palliative treatment BUT pain improvement is observed in 60% to 80%. Combination of hyperthermia (HT) with radiation is strongly compelling. MR is providing accurate, tissue-independent thermometry for intra-procedural guidance of thermal therapy. In this project we aim to combine in an adjuvant setting mild hyperthermia to EBRT for sustained relief of pain in patients with symptomatic bone metastases.

DETAILED DESCRIPTION:
Metastatic disease to the bone is a common cause of pain and other significant symptoms with a detrimental impact into quality of life. Up to 85% of the patients dying from breast, prostate, or lung cancer present bone metastases. External beam radiation therapy (EBRT) is one of the standard palliative treatment modalities effective in palliating painful bone metastases. Using patient-based evaluation method, pain improvement is observed in 60% to 80% of the patients, with 15% to 40% complete pain relief. Combination of hyperthermia (HT) with radiation is strongly compelling as it is based on principles of classic radiobiology, molecular biology, and tumor physiology. Elevating temperature to a supra-physiological level (between 41° and 43°) shows a complementary action when combined with RT with regard to cell killing. Magnetic resonance (MR) imaging is commonly used in clinical routine for radiological diagnostic and staging. Moreover, MR is providing accurate, tissue-independent thermometry for intra-procedural guidance of thermal therapy. In this project we aim to combine in an adjuvant setting mild hyperthermia to EBRT for sustained relief of pain in patients with symptomatic bone metastases. Ex vivo studies for the adaptation of existing MR-guided focused ultrasound (MRgFUS) device were already conducted at University Hospitals of Geneva to the current application demonstrating the high accuracy of the technique for mild hyperthermia treatments. A clinical prospective, interventional, single-center pilot feasibility study will be conducted to assess the clinical application of this technique.

Primary objective

1. Accurate control of spatio-temporal pixel-wise MR thermometry (several hundred pixels): spatial homogeneity of temperature elevation within the tumour and inter-patient reproducibility (expected standard deviation of 0.5°C).
2. Safety and patient tolerance: no adverse effects in surrounding bone and soft tissues, compliance with one-day dual treatment during the first month.

Secondary objectives

1. Complete pain response at 28 days after EBRT + HT based on the International Bone Metastases Consensus Endpoint definition.
2. Pain assessment for the worst pain related to the treated lesion using the Brief Pain Inventory score at baseline, at day 1, day 7, and 28 days after treatment after EBRT + hyperthermia.
3. Health-related quality of life evaluated using self-administered EORTC QLQ-C15-PAL and EORTC QLQ-BM22 (bone metastases module) questionnaires at baseline, day 7, and day 28 after EBRT + hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically proven cancer;

  * cancer-related pain corresponding to a site (or sites) of radiologically confirmed bone metastases with a severity score of at least 2 out of 10 according to the Brief Pain Inventory (NRS scale);
  * age ≥ 18 years;
  * indication for a palliative course of EBRT;
  * osteolytic or mixed (osteoblastic/osteolytic) bone metastases ≤ 5 cm in the largest diameter; target tumours accessibility for device (ribs, extremities, pelvis, shoulders or posterior aspects of spinal vertebra) and at least 1 cm from skin and major nerve bundles;

Exclusion Criteria:

* Inability to provide a written informed consent;
* Karnofsky performance status (KPS) < 60; presence of clinical or radiological evidence of spinal cord compression, a pathological fracture, or an impending fracture needing surgical fixation;
* previous EBRT to study site (or sites);
* participation in another clinical trial and any concurrent treatment with any investigational drug within 4 weeks prior to trial entry;
* inability to comply with study and follow up procedures;
* patients having metal implants, pacemakers or clustered markers non-MR compatible

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Accurate elevation of temperature measured by MRI thermometry (degree celsius) | day 1
  Accurate control of spatio-temporal pixel-wise MR thermometry (several hundred pixels): spatial homogeneity of temperature elevation within the tumour and inter-patient reproducibility (expected standard deviation of 0.5°C).
Safety and patient tolerance according to The adverse events (CTCAE v5.0) (Art. 2 Abs 58 MDR) | day 1
  Safety and patient tolerance: no adverse effects in surrounding bone and soft tissues, compliance with one-day dual treatment during the first month.
  Dermatitis of grade 3 or more - Pain of skin grade 3
  * Skin atrophy grade 3
  * Localized edema of grade 3
  * Bone fracture of grade 3 or more

SECONDARY OUTCOMES:
Complete pain response according to International Bone Metastases Consensus Endpoint score (BPI score) | at 28 days after EBRT + HT
  Complete pain response based on the International Bone Metastases Consensus Endpoint definition.
Pain assessment using Brief Pain Inventory score (BPI score) | at day 1, day 7, and 28 days after treatment after EBRT + hyperthermia.
  Pain assessment for the worst pain related to the treated lesion using the Brief Pain Inventory score
quality of life using EORTC QLQ-C15-PAL (bone metastases module) questionnaires. | day 1, day 7, and 28 days after EBRT + hyperthermia.
  Health-related quality of life evaluated using self-administered EORTC QLQ-C15-PAL (bone metastases module) questionnaires
quality of life using EORTC QLQ-BM22 (bone metastases module) questionnaires. | day 7, and day 28 after EBRT + hyperthermia.
  Health-related quality of life evaluated using self-administered EORTC QLQ-BM22 (bone metastases module) questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided